CLINICAL TRIAL: NCT05240521
Title: A Double-Blind, Placebo-Controlled, Crossover-Over Clinical Trial Investigating the Efficacy and Safety, Tolerability of GA-AT0119 in the Treatment of Irritable Bowel Syndrome With Constipation (IBS-C)
Brief Title: Efficacy and Safety, Tolerability of GA-AT0119 in IBS-C
Acronym: RELAX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Devintec Sagl (Industry)
Collaborators: CEBIS International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CBSDEV21072020
Record Dates: First submitted 2022-01-17; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Irritable Bowel Syndrome With Constipation (IBS-C)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A: GA-AT0119 / Placebo (Other): Cross-over Study
  Interventions: Other: ARM A; Other: ARM B
- ARM B: Placebo / GA-AT0119 (Other): Cross-over Study
  Interventions: Other: ARM A; Other: ARM B

INTERVENTIONS:
Other: ARM A — 30 IBS-C patients will receive GA-AT0119 for 28 days, followed by a washout period of 28 days and Placebo for another 28 days
Other: ARM B — 30 IBS-C patients will receive Placebo for 28 days, followed by a washout period of 28 days and GA-AT0119 for another 28 days

SUMMARY:
Irritable bowel syndrome (IBS) is a common functional bowel disorder that imposes a considerable burden on health-related quality of life (QOL) worldwide. Irritable Bowel Syndrome (IBS) is a common digestive disorder affecting 7-21% of the general population. IBS with predominant constipation (IBS-C) is a subtype of IBS that accounts for more than a third of the IBS diagnosed.

The study Sponsor, Devintec SAGL, presents GA-AT0119, which acts by forming a mechanical barrier on the intestinal mucosa thanks to xyloglucan and pea proteins avoiding the increased intestinal permeability, bacterial invasion to intestinal tissues, and subsequent intestinal inflammation. The formulation of GA-AT0119 is completed with chia seed powder which provides a laxative effect by retaining water in the intestine increasing stool bulk and accelerating fecal transit.

There is increasing evidence that the pathophysiology of IBS is multifaceted involving mucosal inflammation, visceral hypersensitivity, microbial dysbiosis, dietary factors, and altered intestinal permeability (IP). Several studies have shown increased intestinal permeability in patients with irritable bowel syndrome. Serum zonulin, a biomarker of impaired increased permeability, is increased in patients' constipation-predominant irritable bowel syndrome compared to a healthy population and the levels are comparable to celiac disease.

DETAILED DESCRIPTION:
Each subject will be asked to sign the Informed Consent Form (ICF). The patients diagnosed with IBS-C will be randomized in 1:1 ratio. The treatment will be administrated according to the approved leaflet and study procedures. Eligible patients will be randomized to receive either GA-AT0119 or Placebo. Patients will be treated according to the approved leaflet. The study subjects will return at day 7, 15 and day 28 for evaluation. Each subject will undergo a washout period of 28 days. At Day 56 each subject will be evaluated and will receive the crossover therapy line and start administration. Subject will be evaluated at Day 84 at the end of the crossover period. Patients will be evaluated for constipation symptoms, global assessment for tolerability, safety. Each subject will receive a diary where bowel frequency, type and transit time will be completed during product administration. From visit 2 to visit 6, patients will be evaluated for treatment adherence and clinical symptoms recurrences. Each subject will complete 2 additional phone follow-ups Visit for safety reporting and clinical symptoms recurrences according to protocol. During the follow-up visits subject will be evaluated also by using Likert scale for Abdominal Pain and discomfort, Sickness Impact Profile score, IBS-VAS scale and IBS-QoL.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects over 18 years old;
* Subject willing to sign the informed consent;
* The ability to comply with study visits;
* Patients with constipation following diagnostic of IBS-C (Subtypes prevalent presentation of stool in IBS according to the Rome IV Criteria: IBS with constipation (IBS-C) - ( >25% hard stools and <25% loose stools)

Exclusion Criteria:

* Use of gelatin tannate, diosmectite, probiotics, racecadotril or any other drugs or medical devices known to alter gastrointestinal motility or secretion within four weeks prior to enrolment
* Chronic diarrhea caused by cystic fibrosis, coeliac disease, food allergy, diabetes Chronic diarrhea caused by lactose, fructose, or sorbitol intolerance
* Diagnostic of IBS-D
* Use of prebiotics, fiber supplements, laxatives, 5-HT4 agonists, antispasmodic, antidepressants with 4 weeks prior study Baseline visit
* Immunodeficiencies
* Abnormal thyroid function, a history of alcohol abuse or binge drinking, pancreatitis, sphincter of Oddi dysfunction, cholecystitis within the past 6 months, or known allergy to any of the components of the product or placebo
* The patient is a member of the investigational team or his/her immediate family
* Pregnant or breast-feeding women or women planning to become pregnant or breastfeed during the study
* Hypersensitivity to any of the ingredients of the study agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Subjective Symptom Improvement assessed through Likert scale (Discomfort, Bloating Abdominal Pain) at day 7, 15, 28, 56, 84,114,144 | 144 days
  The clinical symptoms that are going to be assessed through the 7 point Likert Scale are: Bloating, Discomfort, abdominal pain.
  Likert scale - level of acceptability:
  1. - Totally unacceptable
  2. - Unacceptable
  3. - Slightly unacceptable
  4. - Neutral
  5. - Slightly acceptable
  6. - Acceptable
  7. - Perfectly Acceptable
Change from baseline in BMI assessed at Day 7,15, 28, 56,84 | 84 days
  The BMI will be evaluated
Change from baseline in stool consistency will be assessed at Day 0, 7, 15, 28, 56, 84, 114, 144, through the Bristol Stool Scale. | 144 days
  Type of stool will be assessed according to the Bristol Stool Chart ((Stool Type 1 - severe constipation, Stool Type 2 - mild constipation, Stool Type 3 - normal, Stool Type 4 - normal, Stool Type 5 - lacking fiber, Stool Type 6 - mild diarrhea, Stool Type 6 - severe diarrhea)
Change from baseline score in IBS-QoL questionnaire (Information Sheet on the Irritable Bowel Syndrome - Quality of Life Measure) at Day 7, 15, Day 28 and Day 56, Day 84, Day 114, Day 144 | 144 days
  Patients will respond to the IBS-QoL questionnaire. The individual responses to the 34 items are summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life.
Change of Sickness Impact Profile score from Baseline to Day 28 and day 56, day 84, Day 114, Day 144 | 144 days
  The generic health status, the physical, mental and social aspects of health-related functioning and behavior aspectes will be measred through - The Sickness Impact Profile (All the items are scored dichotomously (no=0, yes=1); The items reported as "yes" are used to calculate the scores; higher scores indicate more health-related behavioral problems)
Change from Baseline (Day 0) to Day 7, 15, 28, 56 in Zonuline test | 56 days
  Serum Zonuline test will be performed
Change from Baseline Day 0 to Day 7 in the VAS-IBS questionnaire (Visual Analogue Scale for Irritable Bowel Syndrome) evaluated by Patient Journal Daily on each symptom | 7 days
  The VAS-IBS will be assessed through the Patient Journal. In the VAS-IBS the patients record the overall severity of each item on a 100 points line (very severe discomfort = 0 to no discomfort at all = 100).
Change from Baseline Day 0 to Day 7 in the VAS-IBS questionnaire (The Visual Analogue Scale for Irritable Bowel Syndrome) evaluated by Investigator at Day 15, Day 28 and Day 56, Day 84, Day 114, Day 144 | 144 days
  The Investigator will assess the symptoms in patients suffering from IBS - using the Visual Analogue Scale for Irritable Bowel Syndrome (VAS-IBS) questionnaire. In the VAS-IBS the patients record the overall severity of each item on a 100 points line (very severe discomfort = 0 to no discomfort at all = 100).
Number of AE occurrence | 144 days
  Adverse events will be monitored during all the visits till the end of the study and reported accordingly
% of participants with withdrawal due to AE | 144 days
  Withdrawal due to adverse events will be monitored during all the visits till the end of the study and reported accordingly.
Change from baseline in waist circumference assessed at Day 7,15, 28, 56,84 | 84 days
  The waist circumference will be evaluated
Change from baseline in number of stools will be assessed at Day 0, 7, 15, 28, 56, 84, 114, 144 | 144 days
  Number of stools will be assessed

CONTACTS AND LOCATIONS:
Locations (3):
- Bulgaria (3):
  - Outpatient clinic for individual practice for primary medical care Dr. Elenski EOOD, Plovdiv
  - Medical Center Prolet EOOD, Rousse
  - Ambulatory Practice for Primary Outpatient Medical Care SANA OOD, Sofia

IPD SHARING:
Plan to Share IPD: No